CLINICAL TRIAL: NCT07255989
Title: A Study About the Role of Gut Microbiome in Fatty Liver -Fatty Pancreas and Heart Diseases .
Brief Title: Diagnosis of Fatty Pancreas by FibroScan
Acronym: FattyPancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Prof.Reda Mohamed Elbadawy, professor Hepatology , Gastroenterology, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEPHENo5145,2022,BU.; Ministry of Higher education (Other: Benha University)
Record Dates: First submitted 2025-11-17; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: To Assess Feasibility of the New Application
Keywords: Fatty Pancreas , FibroScan

STUDY DESIGN:
Intervention Model Description: Evaluation of uses FibroScan as non invasive method for diagnosis of fatty pancreas
Masking Description: As we are care to early diagnosis of fatty pancreas by simple non invasive method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the patients evaluated clinically , physically and interview after that examination done by Fibr (Experimental)
  Interventions: Device: meeting about the nutrition

INTERVENTIONS:
Device: meeting about the nutrition — In the meeting time abou the nutrition we talk about our ancient egyptian food which confirmed with Carton already present at center of excellence ,

SUMMARY:
Example 2: Interventional study The goal of this observational study is to learn know about the use of FibroScan in diagnosis of fatty pancreas in obese and non obese patients which done for the first time at worldwide as well as Egypt .The participtants already came to do liver FibroScan at center of excellence , Benha University , Egypt. Untill now the diagnosis of fatty pancreas by MRI which accurate and specific and diagnose fatty pancreasif it is more than 6.2% . lough the use of abdominal ultrasound also is proved . The use of digital fibroscan which is easy non invasive , unique as well as we can diagnose fibrosis too in the same sitting .So it is highly recommended to be add with examination of liver by fibroscan.

DETAILED DESCRIPTION:
This Interventional study done for subjects attend Center of excellence , at Benha University . aged of patients was from 30 years to 70 years old , both male and females , obese or non and DM or non . the patients came to do fibroscan to liver . Lab investigations in the form of CBC ,ESR , liver function tests , kidney function tests. Complete lipid profile , HbA1c .clincal and physical examinations done as regard BMI, past history for metabolic diseases , operations and blood transfusion. FibroScan done first to liver while the patients fastinf at least 3 hours with the know specific position recommendation (banana like ).The position for pancreas examination by fibroScan differe as the patient dorsal position/ recumbancy and his hand behind his head . take deep breah and slighlty keep it . some tilting to the left or right . the probe of fibroscan in the epigastrium under the left rib.which totally differe than liver which in the RT anterior axillary line 8 th intercostal space.picture taken , the unique , novality of this modility is the diagnosis of fibrosis too like liver.Grading of aftty pancreas was done as well as fibrosis of pancreas as follow :S1 =264 dB/m , S2 =276 dB/m and S3 =336 dB/m .

ELIGIBILITY:
Inclusion Criteria:

- Subjects aged from 30 to 70 years old , both male and females , DM or not obese or non obese

Exclusion Criteria:

* Exclusion Criteria:

  1. Subjects with significant amount of alcohol consumption or history of alcohol consumption (>60 g/day).
  2. History of steatogenic medications (amiodarone, valproic acid, corticosteroids, tetracyclines).
  3. Patients with a previous history of pancreatic disease

     -

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
prevelance of fatty pancreas 60% which is more common than the expection | 6 months
  the need to raise uo the importance to use FibroScan to diagnosis of fatty pancreas which is novel , unique and invasive , specific

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University , Egypt, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
because the property of the technique

REFERENCES:
- See also: Related Info — http://info@bu.edu.eg